CLINICAL TRIAL: NCT00507806
Title: Microbubble-Enhanced Clotbust Treatment of Acute Ischemic Stroke
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: for administrative reasons
Sponsor: ImaRx Therapeutics (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MRX-815-401
Record Dates: First submitted 2007-07-25; First posted 2007-07-27 (Estimated); Last update posted 2007-07-27 (Estimated); Status verified 2007-07

CONDITIONS: Acute Ischemic Stroke
Keywords: Acute Ischemic Stroke; Microbubbles; Transcranial Doppler ultrasound; TIBI; Symptomatic Intracranial Hemorrhage; modified Rankin Scale; Recanalization; Perflutren
MeSH Terms: conditions — Ischemic Stroke | interventions — perflutren

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: perflutren lipid microsphere
  Other Names: Definity

SUMMARY:
The study is designed to examine the safety, tolerability, and activity of a combination of microbubbles (perflutren lipid microsphere [Definity®]) and continuous monitoring with 2 MHz transcranial Doppler ultrasound (TCD) as an adjunctive therapy to tissue plasminogen activator (tPA) treatment in subjects with acute ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

* Measurable focal neurological deficit (National Institutes of Health Stroke Scale [NIHSS] score > 4 points)
* tPA eligible
* Occlusion of the middle cerebral artery

Exclusion Criteria:

* Right to left cardiac shunt
* Uncontrolled hypertension
* Absent temporal windows

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2005-03; Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Incidence of symptomatic intracranial hemorrhage | 72 hours

SECONDARY OUTCOMES:
Complete recanalization of the occluded artery (TIBI 4-5) | End of treatment
NIHSS score of 0-2 | 24 hours
Favorable outcome (modified Rankin Scale or NIHSS 0-1) | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Andrei Alexandrov, MD, Principal Investigator — The University of Texas Health Science Center, Houston

REFERENCES:
- [Background] Alexandrov AV, Molina CA, Grotta JC, Garami Z, Ford SR, Alvarez-Sabin J, Montaner J, Saqqur M, Demchuk AM, Moye LA, Hill MD, Wojner AW; CLOTBUST Investigators. Ultrasound-enhanced systemic thrombolysis for acute ischemic stroke. N Engl J Med. 2004 Nov 18;351(21):2170-8. doi: 10.1056/NEJMoa041175. PMID 15548777